CLINICAL TRIAL: NCT02202135
Title: A Phase III, Multicentre, Randomised, Double-Blind Comparative Study to Evaluate the Efficacy and Safety of Ceftaroline Fosamil (600 mg Every 8 Hours) vs Vancomycin Plus Aztreonam in the Treatment of Patients With Complicated Bacterial Skin and Soft Tissue Infections With Evidence of Systemic Inflammatory Response or Underlying Comorbidities.
Brief Title: Evaluation of Ceftaroline Fosamil vs Vancomycin Plus Aztreonam in the Treatment of Patients With Skin Infections.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Overall study status is changed to "Terminated" due to low enrollment
Sponsor: Pfizer (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D3720C00001sub
Record Dates: First submitted 2014-07-25; First posted 2014-07-28 (Estimated); Results first posted 2016-03-31 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Complicated Skin and Soft Tissue Infection
Keywords: complicated skin and soft tissue infections (cSSTI); skin infection; ceftaroline; wound infection; cellulitis; burn infection; bacterial infection; vancomycin
MeSH Terms: conditions — Soft Tissue Infections; Cellulitis; Wound Infection; Bacterial Infections | interventions — Ceftaroline; Vancomycin; Aztreonam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ceftaroline fosamil (Experimental): Patients will receive 600 mg of ceftaroline fosamil administered as a 120-minute intravenous infusion very 8 hours. Each dose will be infused in a volume of 250 mL over 120-minutes followed by aztreonam placebo in a volume of 100 mL infused over 30 minutes every 8 hours. In addition vancomycin placebo will be given in a volume of 250 mL infused over 120 minutes every 12 hours. Doses will be adjusted according to the patient's renal function.
  Interventions: Drug: Ceftaroline fosamil
- Vancomycin plus aztreonam (Active Comparator): Patients will receive combination of vancomycin plus aztreonam. Dose of vancomycin will be based on the patient's actual weight and will receive intravenous vancomycin every 12 hours with each dose infused over 120-minutes. Aztreonam dose will be 1 gram intravenously in a volume of 100 mL infused over 30 minutes every 8 hours. In addition, ceftaroline fosamil placebo will be given in a volume of 250 mL infused over 120 minutes every 8 hours. Doses adjusted according to patients renal function
  Interventions: Drug: Vancomycin; Drug: Aztreonam

INTERVENTIONS:
Drug: Ceftaroline fosamil — IV ceftaroline 600mg every 8 hours
  Arms: Ceftaroline fosamil
Drug: Vancomycin — IV vancomycin 15mg/kg every 12 hours
  Arms: Vancomycin plus aztreonam
Drug: Aztreonam — IV aztreonam 1 g every 8 hours
  Arms: Vancomycin plus aztreonam

SUMMARY:
The purpose of this study is to evaluate the effects of Ceftaroline Fosamil versus Vancomycin plus Aztreonam in treatment of patients with complicated bacterial skin and soft tissue infections.

DETAILED DESCRIPTION:
A Phase III, Multicentre, Randomised, Double-Blind Comparative Study to Evaluate the Efficacy and Safety of Ceftaroline Fosamil (600 mg every 8 hours) Versus Vancomycin Plus Aztreonam in the Treatment of Patients with Complicated Bacterial Skin and Soft Tissue Infections With Evidence of Systemic Inflammatory Response or Underlying Comorbidities

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older - Complicated skin and skin structure infection (cSSTI) - Infection of sufficient severity to warrant hospitalization - Infection of sufficient severity such that it is expected to require at least 5 days of intravenous antibiotic therapy. patients must have a positive culture for MRSA that has been obtained from the skin infection site and/or blood samples at any time within the 72hrs before the first dose.

Exclusion Criteria:

* Received systemic antibacterial drugs for greater than 24 hours within 96 hours prior to first dose of study drug - Uncomplicated skin and skin structure infections, skin infections suspected to be caused by viral or fungal pathogens - Diabetic foot infections, decubitus ulcers, ulcers due to peripheral vascular disease - Infection caused by human or animal bites, sternal wound infections, bone infection or arthritis due to an infection, critical limb ischemia of the affected limb - Chronic liver disease or severe impaired renal function, severe low white blood cell count, burns on greater than 15% of total body surface area, necrotizing skin infection, amputation required of primary site of infection, sustained shock

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MSD, Study Director — AstraZeneca
Locations (22):
- Research site, Córdoba, Argentina
- Brazil (3):
  - Research site, Salvador, Estado de Bahia
  - Research site, Passo Fundo, Rio Grande do Sul
  - Research site, São José do Rio Preto
- Research site, Pleven, Bulgaria
- Research site, Temuco, Chile
- Research site, Zagreb, Croatia
- Research site, Athens, Greece
- Israel (4):
  - Research site, Haifa
  - Research site, Ramat Gan
  - Research site, Safed
  - Research site, Tel Aviv
- Research site, Milan, Italy
- Research site, Lodz, Poland
- Research site, Bucharest, Romania
- South Africa (2):
  - Research site, Dundee
  - Research site, Worcester
- Spain (2):
  - Research site, Granada
  - Research site, Terrassa
- Turkey (Türkiye) (3):
  - Research site, Ankara
  - Research site, Diyarbakır
  - Research site, Izmir

REFERENCES:
- [Derived] Dryden M, Zhang Y, Wilson D, Iaconis JP, Gonzalez J. A Phase III, randomized, controlled, non-inferiority trial of ceftaroline fosamil 600 mg every 8 h versus vancomycin plus aztreonam in patients with complicated skin and soft tissue infection with systemic inflammatory response or underlying comorbidities. J Antimicrob Chemother. 2016 Dec;71(12):3575-3584. doi: 10.1093/jac/dkw333. Epub 2016 Sep 1. PMID 27585969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 4 patients were enrolled from 2 centres in 1 regions in this study. The first patient was enrolled on 15 September 2014 and the last patient last visit was on 02 January 2015.
Groups:
- Ceftaroline: Ceftaroline fosamil 600 mg 120 min
Period: Overall Study
Arm/Group | Ceftaroline
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Randomized patients
Arm/Group | Ceftaroline
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.25 (4.875)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response at TOC
Description: Clinical cure is defined as resolution or improvement of signs and symptoms compared to baseline and no further antimicrobial therapy is necessary. Clinical failure is defined as any of the following: persistence or worsening in signs or symptoms, or requirement for concomitant antibiotic therapy, or requirement of an unplanned surgical intervention >48 hours after the first dose, or death caused by skin infection, or an AE leading to study drug discontinuation with alternative antimicrobial therapy required, or diagnosis of osteomyelitis >=8 days after the first dose.
Time Frame: 7 to 20 days after last dose of study drug
Population: Randomized
Measure: Number; unit: Participant
Arm/Group | Ceftaroline
Number analyzed (Participants) | 4
Participant
  Clinical cure | 3
  Clinical failure | 0
  Indeterminate | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of the first dose of study drug up to TOC visit (8 to 15 days after the last dose). Serious AEs were collected from time of signature of informed consent up to the LFU visit (21 to 35 days after the last dose).
Arm/Group | Ceftaroline
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline (N=4)
Pneumonia (Infections and infestations) | 1 (1) — SAE started at 12:00 pm on and resolved at 13:00 pm on 2014-08-08. It was reported as important medical event which was assessed as moderate and unrelated to study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline (N=4)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Urinary tract (Infections and infestations) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to use such Confidential study information and not to disclose them to any other third parties, except that the undersigned shall not be prevented from using or disclosing information: (a) which by written records was previously known; (b) which is now public knowledge, (c) which is lawfully obtained by the undersigned from sources who have a lawful right to disclose such information.